CLINICAL TRIAL: NCT03160222
Title: Validation of Bedside Ultrasound to Predict Body Composition in Non- and Critically Ill Patients: The USVALID Prospective Study
Brief Title: Validation of Bedside Ultrasound to Predict Body Composition in Non- and Critically Ill Patients
Acronym: USVALID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Arabella Fischer, MD, Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1848/2016
Record Dates: First submitted 2016-12-30; First posted 2017-05-19 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Ultrasound; Body Composition
Keywords: reliability; bioelectrical impedance analysis; computed tomography; strength; mobility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Body Composition Measurements (Other): Body composition measurements comprise the ultrasound measurement of fat and muscle thickness of both upper arms and thighs, the bioelectrical impedance analysis (BIA), measurement of weight, handgrip strength, overall muscle strength (Medical Research Council scale) and questionnaires about physical activity, nutrition and fluid status.
  Interventions: Other: Body Composition Measurements

INTERVENTIONS:
Other: Body Composition Measurements — Body composition measurements comprise the ultrasound measurement of fat and muscle thickness of both upper arms and thighs, the bioelectrical impedance analysis (BIA), measurement of weight, handgrip strength, overall muscle strength (Medical Research Council scale) and questionnaires about physical activity, nutrition and fluid status.

SUMMARY:
The prospective study will include 200 patients and 50 critically ill patients, who had an abdominal computed tomography (CT) scan including the L3 level for any clinical reason. Ultrasound scans of the anterior thighs and forearms will be taken after the CT scan within 48 hours. Bioelectrical impedance analysis (BIA) will also be performed. In addition muscle strength, mobility, physical function and nutrition will be assessed. Primary outcome is the prediction of CT-based whole body muscle and fat volume and BIA-based fat and lean body mass from ultrasound-based muscle and fat thickness. Other secondary outcomes include the intra- and interrater reliability of the CT evaluation and ultrasound examination of muscle and fat mass. The relationship between clinical aspects (strength, mobility, physical function, nutrition) and whole body composition is another secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* cross-sectional abdominal CT scan including the level of L3 vertebra for any clinical reason
* study-related ultrasound examination must take place within 48 hours of CT

Exclusion Criteria:

* patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-01; Primary Completion 2019-03-22 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
prediction (r2) of CT-based whole body muscle volume from ultrasound-based muscle thickness | Ultrasound measurement once-only within 48 hours after the CT scan
  In a linear regression model, the dependent variable is CT-based whole body muscle volume. The independent variable is ultrasound-based muscle thickness. The prediction (r2) of CT-based muscle volume in the multiple linear regression model is the outcome.
prediction (r2) of CT-based whole body fat volume from ultrasound-based fat thickness | Ultrasound measurement once-only within 48 hours after the CT scan
  In a linear regression model, the dependent variable is CT-based whole body fat volume. The independent variable is ultrasound-based fat thickness. The prediction (r2) of CT-based fat volume in the multiple linear regression model is the outcome.

SECONDARY OUTCOMES:
prediction (r2) of BIA-based whole body muscle volume from ultrasound-based muscle thickness | BIA measurement once-only within 48 hours after the CT scan
  In a linear regression model, the dependent variable is BIA-based whole body muscle volume. The independent variable is ultrasound-based muscle thickness. The prediction (r2) of BIA-based muscle volume in the multiple linear regression model is the outcome.
prediction (r2) of BIA-based whole body fat volume from ultrasound-based fat thickness | BIA measurement once-only within 48 hours after the CT scan
  In a linear regression model, the dependent variable is BIA-based whole body fat volume. The independent variable is ultrasound-based fat thickness. The prediction (r2) of BIA-based fat volume in the multiple linear regression model is the outcome.
intrarater reliability (bias in Bland Altman analysis) of ultrasound muscle/fat thickness | repeated US measurement in 60 patients once-only within 48 hours after the CT scan
  For intrarater reliability each of the 5 examiners repeats the ultrasound measurement in 12 patients. In a Bland Altman analysis, the mean difference (=bias) in muscle/fat thickness between repeated measurements of the same examiner is the outcome.
interrater reliability (bias in Bland Altman analysis) of ultrasound muscle/fat thickness | repeated US measurement in 60 patients once-only within 48 hours after the CT scan
  For interrater reliability each of the 10 different pairs of examiners analyzes 6 patients. For each pair both examiners perform the ultrasound examination. In a Bland Altman analysis, the mean difference (=bias) in ultrasound muscle/fat thickness between examiners is the outcome.
muscle strength in patients with different CT-based body compositions (sarcopenia, malnutrition, obesity, sarcopenic obesity) | muscle strength measurement once-only within 48 hours after the CT scan
  Muscle strength is measured with MRC scale and hand dynamometry. The outcome is muscle strength evaluated in different patient's group according to their CT-based body composition. Sarcopenia is defined as lowered L3 skeletal muscle index. Malnutrition is defined at a BMI beneath18,5 kg/m². Obesity is defined as a BMI above or equal to 30 kg/m². Sarcopenia obesity is defined as lowered L3 skeletal muscle indices and a BMI above or equal to 30 kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Arabella Fischer, Dr., Principal Investigator — Medical University of Vienna; Michael Hiesmayr, Prof. Dr., Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen W, Punyanitya M, Wang Z, Gallagher D, St-Onge MP, Albu J, Heymsfield SB, Heshka S. Visceral adipose tissue: relations between single-slice areas and total volume. Am J Clin Nutr. 2004 Aug;80(2):271-8. doi: 10.1093/ajcn/80.2.271. PMID 15277145
- [Background] Sanada K, Kearns CF, Midorikawa T, Abe T. Prediction and validation of total and regional skeletal muscle mass by ultrasound in Japanese adults. Eur J Appl Physiol. 2006 Jan;96(1):24-31. doi: 10.1007/s00421-005-0061-0. Epub 2005 Oct 19. PMID 16235068
- [Background] Weijs PJ, Looijaard WG, Dekker IM, Stapel SN, Girbes AR, Oudemans-van Straaten HM, Beishuizen A. Low skeletal muscle area is a risk factor for mortality in mechanically ventilated critically ill patients. Crit Care. 2014 Jan 13;18(2):R12. doi: 10.1186/cc13189. PMID 24410863
- [Background] Paris MT, Mourtzakis M, Day A, Leung R, Watharkar S, Kozar R, Earthman C, Kuchnia A, Dhaliwal R, Moisey L, Compher C, Martin N, Nicolo M, White T, Roosevelt H, Peterson S, Heyland DK. Validation of Bedside Ultrasound of Muscle Layer Thickness of the Quadriceps in the Critically Ill Patient (VALIDUM Study). JPEN J Parenter Enteral Nutr. 2017 Feb;41(2):171-180. doi: 10.1177/0148607116637852. Epub 2016 Jul 11. PMID 26962061
- [Background] Prado CM, Heymsfield SB. Lean tissue imaging: a new era for nutritional assessment and intervention. JPEN J Parenter Enteral Nutr. 2014 Nov;38(8):940-53. doi: 10.1177/0148607114550189. Epub 2014 Sep 19. PMID 25239112
- [Background] Takai Y, Ohta M, Akagi R, Kato E, Wakahara T, Kawakami Y, Fukunaga T, Kanehisa H. Applicability of ultrasound muscle thickness measurements for predicting fat-free mass in elderly population. J Nutr Health Aging. 2014;18(6):579-85. doi: 10.1007/s12603-013-0419-7. PMID 24950147